CLINICAL TRIAL: NCT00420043
Title: A Phase I, Two Arm, Open-label, Randomized, Study to Investigate the Effect of Food on the Bioavailability of a Single 800 mg Imatinib Dose in Modified Release Formulations (MR3 and MR4) and Compare the Bioavailability Between MR3, MR4 and Imatinib 400 mg Twice Daily Immediate Release Tablet (IR) in Healthy Subjects
Brief Title: Effect of Food on Bioavailability of Modified Release Formulations of Imatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571O2103
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Food effect; bioavailability; pharmacokinetic; STI571; modified release formulation of STI571; CML; Chronic Myeloid Leukemia; Philadelphia Chromosome; imatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- imatinib 800mg (Experimental)
  Interventions: Drug: imatinib
- imatinib 400mg (Active Comparator)
  Interventions: Drug: imatinib

INTERVENTIONS:
Drug: imatinib
  Other Names: STI571

SUMMARY:
This study will evaluate the effect of food on the relative bioavailability of a single dose of imatinib given as a 800 mg modified release tablet, compared to twice-daily doses of 400 mg film-coated tablets. There will be a 8 day wash out phase between treatments and a 1 week safety period at the end of the study. Each participant will receive all four treatments.

ELIGIBILITY:
Inclusion criteria

* Healthy male or female subjects (postmenopausal women), 18-65 years of age
* Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion criteria

* Smokers within 3 months
* Subjects using any prescription drug or over-the-counter (OTC) medication (including herbal and alternative medication) within 3 weeks prior to dosing.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* A past medical history or presence of clinically significant ECG abnormalities
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* History of medications pre-disposing the subjects for GI bleedings/cerebral hemorrhage.
* Women taking any biphosphonates (Fosomax like drugs)
* History of being immunocompromised, including a positive HIV test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* Females nursing infants. Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To compare the bioavailability of Modified Release formulations to 400 mg immediate release (IR) tablet when administered twice-daily (both given with a low fat meal).

SECONDARY OUTCOMES:
To compare the relative bioavailability of a single daily 800 mg dose of modified release formulations with a high fat meal and a low fat (regular) meal, to modified release formulations after over-night fasting in healthy volunteers.
To compare safety and tolerability of the 800 mg daily dose modified release formulations with or without food

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis